CLINICAL TRIAL: NCT00802893
Title: Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation, Parallel Study of Oral 6R-BH4 in Subjects With Isolated Systolic Hypertension and Endothelial Dysfunction
Brief Title: Oral 6R-BH4 for the Treatment of Isolated Systolic Hypertension and Endothelial Dysfunction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: We were unable to recruit any subjects into this study so no subjects completed the protocol. Therefore, we are unable to provide any conclusions.
Sponsor: Johns Hopkins University (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00014296
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Isolated Systolic Hypertension; Endothelial Dysfunction
Keywords: Isolated Systolic Hypertension with Endothelial Dysfunction
MeSH Terms: conditions — Isolated Systolic Hypertension | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Drug (Experimental)
  Interventions: Drug: 6R-BH4
- Placebo Comparator (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 6R-BH4 — 6R-BH4 5mg/kg or Placebo BID for four weeks and then 8 week dose-escalation period
  Arms: Experimental Drug
Other: Placebo — placebo given BID for entire length of study
  Arms: Placebo Comparator

SUMMARY:
This study is designed to assess the safety and efficacy of twice-daily oral dosing of 6R-BH4 to improve endothelial function, reduce systolic blood pressure and reduce arterial stiffness.

DETAILED DESCRIPTION:
By comparing values measured at different timepoints, the study is expected to provide insight regarding the ability of 6R-BH4, administered along with their currently prescribed antihypertension medications, to improve endothelial function, reduce SBP, and reduce arterial stiffness in patients with ISH and endothelial dysfunction

ELIGIBILITY:
Inclusion Criteria:

* No change in prescribed antihypertension medications within the previous 30 days
* Study staff able to visualize and measure the brachial artery diameter by high resolution vascular ultrasound required for FMD measurements
* ISH with the following mean seated BP: SBP > 145 and < 180 mmHg. Diastolic blood pressure < 90mmHg

Exclusion Criteria:

* Has known hypersensitivity to 6RBH4 or its excipients
* Pregnant or breastfeeding at screening
* Use of any investigational product or investigational medical device within 30 days prior to screening
* Current disease or condition that would interfere with study participation or safety such as the following: heart failure, atrial fibrillation, aortic valve disease, bleeding disorders, history of repeated syncope or vertigo, severe GERD, GI ulcer, symptomatic coronary or peripheral vascular disease, arrhythmia, serious neurologic disorders including seizures, organ transplant or organ failure
* Hypertension secondary to other medical conditions
* Any severe comorbid condition that would limit life expectancy to <6 months
* Current use of any nicotine containing substances
* History of drug or alcohol abuse
* MI, stroke or surgery within 90 days before Screening Visit
* CABG within 6 months before the Screening Visit
* Serum creatinine >2.0mg/dl or AST, ALT, GGT levels >2times upper limit of normal
* Concomitant treatment with: any drug known to inhibit folate metabolism, any phosphodiesterase-5 or -3 inhibitor
* Previous treatment with any formulation of BH4

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: 6R-BH4: 6R-BH4 5mg/kg or Placebo BID for four weeks and then 8 week dose-escalation period
  OR
  Placebo: placebo given BID for entire length of study
Period: Overall Study
Arm/Group | All Participants
Started | 3
Completed | 0
Not Completed | 3
Not completed — study terminated | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 3
Age, Customized [Count of Participants; unit: Participants]
  >=40, years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Efficacy of 6R-BH4 Versus Placebo to Improve Endothelia Function
Time Frame: 4-6 weeks
Population: Due to difficulties recruiting, this study was terminated and no data was collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Evaluate the Efficacy of Oral 6R-BH4 Versus Dosage-equivalent Placebo to Improve Endothelia Function, to Reduce SBP, to Reduce Arterial Stiffness
Time Frame: 4-8 weeks
Population: Due to difficulties recruiting, this study was terminated and no data was collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Unknown. Due to difficulties recruiting, this study was terminated and no data was collected.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes